CLINICAL TRIAL: NCT05406128
Title: The Effect of Erector Spina Plan Block Application Time on Postoperative Anxiety in Cases of Lumbar Disc Hernioplasty
Brief Title: The Effect of Erector Spina Plan Block Application Time on Postoperative Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, fulya eser, assistant doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: anxiety
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Recovery of Postoperative
Keywords: block timing; quality of recovery; erector spina plan block

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative group (Active Comparator): Erector spina plane block will be applied to preoperative group patients in the preoperative period.
  Interventions: Other: preoperative erector spina plane block
- intraoperative group (Active Comparator): In the intraoperative group, erector spina plane block will be applied after anesthesia induction.
  Interventions: Other: intraoperative erector spina plane block

INTERVENTIONS:
Other: preoperative erector spina plane block — Erector spina plane block will be applied to preoperative group patients in the preoperative period.
  Arms: preoperative group
Other: intraoperative erector spina plane block — In the intraoperative group, erector spina plane block will be applied after anesthesia induction.
  Arms: intraoperative group

SUMMARY:
we aimed to compare the effect of preoperative awake or post-induction erector spina plane block on patient anxiety and recovery quality in patients who will undergo elective lumbar disc hernioplasty.

DETAILED DESCRIPTION:
Postoperative recovery quality can be tested with the Quality of Recovery-40 (QoR-40) questionnaire. Preoperative anxiety can be detected through structured and standardized screening with the State-Trait Anxiety Inventory (STAI) I and II. In our study, 108 patients between the ages of 18-70 who were planned for lumbar disc hernioplasty will be included. Preoperative Quality of Recovery-40 (QoR40), STAI I and II scores (anxiety questionnaire) will be administered to each patient.The patients will be divided into two groups as preoperative ve intraoperative group. Erector spina plane block will be applied to preoperative group patients in the preoperative period. In the intraoperative group, erector spina plane block will be applied after anesthesia induction. The STAI and Quality of Recovery-40 (QoR40) questionnaire will be repeated postoperatively, the Numerical Rating Scale (NRS) and postoperative patient satisfaction will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* American Society of Anesthesiologists score I-II-III
* Patients who can read and write
* Can speak Turkish language clearly

Exclusion Criteria:

* Visual and hearing impaired
* Those with dementia
* Known serious heart, kidney and liver diseases
* Life-threatening hematological diseases
* Central and peripheral neurological diseases
* Psychiatric disorders
* History of allergy to amide type local anesthetics
* Infection in the block area
* Bleeding diathesis
* Morbidly obese (patients with BMI 40 and above)
* A history of narcotic drug use within 24 hours before the operation
* Those with narcotic substance and alcohol addiction related to chronic pain
* Patients who refused to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-06-07 (Estimated); Primary Completion 2022-09-07 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The quality of postoperative functional recovery (QoR-40) score | 24 hours
  The quality of postoperative functional recovery will assess using the QoR-40, which assesses physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item is rated on a 5-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score ranges from 40 (poorest quality of recovery) to 200 (the best quality of recovery). The QoR-40 will administer one day before surgery in outpatient clinics of anesthesiology, and before discharge from hospital on the first postoperative day.

SECONDARY OUTCOMES:
Spielberg State-Trait Anxiety Inventory (STAI) score | 4 hours
  The test scores between 20 and 80, with higher scores indicating more generalized and stronger anxiety. Preoperative and postoperative STAI I score questions will be asked.
Numerical Rating Scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No